CLINICAL TRIAL: NCT04783207
Title: A Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Effects of Mitopure (Urolithin A) on Skeletal Muscle Function, Iron Metabolism and Endurance Performance in Athletes
Brief Title: Effects of Mitopure (Urolithin A) on Skeletal Muscle Function, Iron Metabolism and Endurance Performance
Acronym: ENDURO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amazentis SA (Industry)
Collaborators: Australian Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 21.01.AMZ/ENDURO
Record Dates: First submitted 2021-02-05; First posted 2021-03-05 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement containing Mitopure (Active Comparator)
  Interventions: Dietary Supplement: Mitopure
- Placebo Supplement (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Mitopure — Softgel containing 250 mg of Urolithin A (Mitopure) with excipients. 4 soft-gels to be taken daily
  Arms: Supplement containing Mitopure
Dietary Supplement: Placebo — Softgel containing only excipients. 4 soft-gels to be taken daily
  Arms: Placebo Supplement

SUMMARY:
This is a randomized, double-blind, placebo-controlled study enrolling 36 (16 Elite and 20 Sub-Elite trained endurance runners (18 placebo and 18 Mitopure intervention) who are 18-40 years of age. Mitopure or Placebo supplement, will be given as a daily oral dose for 4-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-40 years
* Participants will be running >100 km/week
* Elite participants will be required to have a 3,000 m running personal best time below 9:00 (mm:ss), and/or a VO2max result greater than 65 ml·kg-1·min-1
* The sub-elite cohort will have a 3,000 m running personal best faster than 10:00 min and/or a VO2max >60 ml·kg-1·min-1
* Agree to participate in one of two ~4 week training camps been held between March-October 2021.
* Signed informed consent

Exclusion Criteria:

* Subjects with diagnosed medical conditions involving thyroid function or other chronic disturbances of metabolic rate
* Subjects who are unable to complete the training or testing protocols

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Trained elite and sub-elite male runners will participate in a sports training camp
Enrollment: 42 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in plasma levels over time of creatine kinase (CK) | 4 weeks
  Muscle damage and recovery biomarker
Change in race performance time during a 3000 m track race in elite runners | 4-weeks

SECONDARY OUTCOMES:
Change from baseline in aerobic capacity (VO2max) | 4-weeks
Change from baseline in running economy via indirect calorimetry | 4-weeks
Change from baseline in lean body mass via Dual-energy X-ray Absorptiometry (DXA) | 4-weeks
Change from baseline in body fat mass via Dual-energy X-ray Absorptiometry (DXA) | 4-weeks
Change from baseline in Resting Metabolic Rate (RMR) | 4-weeks
Change from baseline in maximal muscle strength during 1-repetition maximum leg press | 4-weeks
change in iron absorption and hemoglobin mass via determination of carboxyhaemoglobin (percent HbCO) | 4-weeks
  only in sub-elite runners
Change in acylcarnitines levels via metabolomics in plasma | 4-weeks
change in mitochondrial function via respirometry in muscle biopsies (sub-elite runners only) | 4-weeks
change in mitochondrial gene expression via RNA-seq in muscle biopsies (sub-elite runners only) | 4-weeks
change in plasma levels of Urolithin A | 4-weeks
change in plasma levels of inflammatory marker CRP | 4-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Louise Burke, OAM PhD, Principal Investigator — Australian Catholic University
Locations (1):
- Australian Catholic University/Australian Institute of Sports, Canberra, Australia

IPD SHARING:
Plan to Share IPD: No